CLINICAL TRIAL: NCT04835168
Title: A Randomized, Placebo-Controlled, Double-Blind, Multicenter Study to Evaluate Safety and Pharmacokinetics of Orodispersible BT-11 in Active Eosinophilic Esophagitis
Brief Title: Safety and Pharmacokinetics of Orodispersible BT-11 in Active Eosinophilic Esophagitis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The closure of the study is driven by the decision to redesign the study protocol for future studies.
Sponsor: NImmune Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BT-11-EoE
Record Dates: First submitted 2021-03-10; First posted 2021-04-08 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BT-11 low (Experimental): Oral
  Interventions: Drug: BT-11 low
- BT-11 high (Experimental): Oral
  Interventions: Drug: BT-11 high
- Placebo (Placebo Comparator): Oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BT-11 low — Oral
  Arms: BT-11 low
Drug: BT-11 high — Oral
  Arms: BT-11 high
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
The proposed Phase 1b study design was a randomized, placebo-controlled, double-blind, study to evaluate the safety and pharmacokinetics of oral BT-11 in active eosinophilic esophagitis.

ELIGIBILITY:
No patients enrolled

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-30 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of AEs | 12 Weeks

IPD SHARING:
Plan to Share IPD: No